CLINICAL TRIAL: NCT05957822
Title: Comparison of Viscoelastic Test-guided and Preemptive Tranexamic Acid Administration Strategies in High-risk Non-cardiac Surgery
Brief Title: Goal-directed vs Preemptive Tranexamic Acid Administration in Non-cardiac Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); Asan Medical Center (Other); Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HI22C195200-1-1
Record Dates: First submitted 2023-07-07; First posted 2023-07-24 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Arthritis Knee; Spine Fusion; Prostate Cancer; Arthritis of Hip; Hepatic Cancer
Keywords: bleeding; viscoelastic test; tranexamic acid; transfusion; thromboembolism; fibrinolysis; seizure
MeSH Terms: conditions — Prostatic Neoplasms; Liver Neoplasms; Hemorrhage; Thromboembolism; Seizures

STUDY DESIGN:
Intervention Model Description: randomized prospective multicenter non-inferior
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TXA empirical (Active Comparator): Empirical Tranexamic acid (TXA) administration after the anesthesia induction
  Interventions: Drug: TXA
- TXA TEG6-triggered (Experimental): When LY30≥3% or MA<54 mm in CRT of TEG6, Tranexamic acid (TXA) is administered
  Interventions: Drug: TXA; Diagnostic Test: TEG6
- TXA TEG6-non-triggered (Experimental): When LY30<3% or MA ≥ 54 mm in CRT of TEG6, Tranexamic acid (TXA) is not administered
  Interventions: Diagnostic Test: TEG6

INTERVENTIONS:
Drug: TXA — Tranexamic acid injection 8-10mg/kg
  Other Names: TXA administration
  Arms: TXA TEG6-triggered; TXA empirical
Diagnostic Test: TEG6 — performing thromboelastography (TEG6)
  Other Names: thromboelastography 6
  Arms: TXA TEG6-non-triggered; TXA TEG6-triggered

SUMMARY:
The present study is a multi-center randomized prospective non-inferiority trial. The study's primary objective is to compare the coagulation profile upon using two different TXA administration strategies: empirical TXA administration vs. viscoelastic test-based goal-directed TXA administration in high-risk non-cardiac surgery. The secondary objectives include comparing the amount of bleeding, incidents of hyper-fibrinolysis, thromboembolic complications, and postoperative seizures. Researchers assumed that goal-directed tranexamic acid (TXA) administration using viscoelastic field tests would not be inferior to the empirical TXA administration strategy in reducing postoperative bleeding and hyper-fibrinolysis. It also would be beneficial in lowering TXA-induced thromboembolic complications and seizures.

DETAILED DESCRIPTION:
The present study is a multi-center randomized prospective placebo-controlled non-inferiority trial. This study's primary objective is to compare the coagulation profile upon using two different TXA administration strategies: empirical TXA administration vs. viscoelastic test-based goal-directed TXA administration in non-cardiac surgery. The secondary objectives include determining the inter-group differences in hyper-fibrinolysis, during postoperative 2bleeding, thromboembolic complications, and postoperative seizures. Researchers hypothesized that goal-directed TXA administration using viscoelastic field tests would not be inferior to the empirical TXA administration strategy in reducing postoperative bleeding and hyper-fibrinolysis. Researchers also expect that goal-directed TXA administration would be beneficial in lowering TXA-induced thromboembolic complications and seizure risks.

ELIGIBILITY:
Inclusion Criteria patients undergoing following surgery

* spinal fusion surgery with more than 2 levels
* total hip arthroplasty
* total knee arthroplasty
* open prostatectomy
* hepatectomy

Exclusion Criteria:

* pregnancy
* refusal of allogenic blood transfusion
* taking thrombin
* history of thromboembolic and familial hypercoagulability disease
* recent history of myocardial infarction or ischemic cerebral infarction (within 90 days)
* hypersensitive to TXA
* histroy of convulsion or epilepsy
* taking hemodialysis
* history of Heparin-induced thrombocytopenia

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
CRT maximal amplitude | 24 hours
  maximal amplitude of CRT test

SECONDARY OUTCOMES:
CK reaction time | 24 hours
  value of r-time of CK test
CK alpha angle | 24 hours
  value of alpha-angle of CK test
CRT maximal lysis | 24 hours
  value of maximal lysis of CRT test
CFF maximal amplitude | 24 hours
  value of maximal amplitude of CFF test
Hemoglobin | 24 hours
  serum hemoglobin value
packed RBC | 6 hours
  number of unit, transfused packed RBC
fresh frozen plasma | 6 hours
  number of unit, transfused fresh frozen plasma
cryoprecipitate | 6 hours
  number of unit, transfused cryoprecipitate
platelet | 6 hours
  number of unit, transfused platelet (apheresis) or platelet concentrate
seizure | 48 hours
  incidence of postoperative seizure
thromboembolism | 48 hours
  incidence of postoperative myocardial infarction, cerebral infarction, pulmonary thrombosis, intestinal infarction
postoperative bleeding | 48 hours
  amount of bleeding from surgical drain
re-operation | 48 hours
  incidence of re-operation due to postoperative bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD, PhD, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes